CLINICAL TRIAL: NCT03633032
Title: Radiation-free Bone Imaging by Ultrashort Echo Time (UTE) Magnetic Resonance Tomography (MRT)
Brief Title: Radiation-free Bone Imaging UTE MRI in Healthy and Diseased Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roman Guggenberger (Other)
Responsible Party: Sponsor-Investigator, Roman Guggenberger, PD Dr. med. Roman Guggenberger, Sponsor-Investigator, Senior Physician, Institute of Diagnostic and Interventional Radiology, University Hospital Zurich, University of Zurich, Switzerland, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USZ_Radiationfree bone imaging
Record Dates: First submitted 2018-07-12; First posted 2018-08-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Bone Anatomy; Bone Diseases
Keywords: bone imaging; MRI; UTE; radiation-free; ultrashort echo time ; anatomy
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Intervention Model Description: Bone anatomy will be compared between different imaging modalities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UTE MRI (Other)
  Interventions: Diagnostic Test: Acquiring of ultrashort echo time (UTE) MRI sequences

INTERVENTIONS:
Diagnostic Test: Acquiring of ultrashort echo time (UTE) MRI sequences — Modern MRI sequences (ultrashort echo time (UTE)) for a better depiction of bone anatomy

SUMMARY:
In summary, the investigators want to investigate whether UTE sequences are capable to replace imaging techniques involving ionizing radiation for bone imaging in the future. This would improve patient care greatly and might reduce medical imaging associated cancer risk drastically from an epidemiological standpoint. This field of research can be considered cutting-edge. The investigators determine this study promising to provide substantial generalizable knowledge and hope that this study results will improve patient care worldwide considerably.

DETAILED DESCRIPTION:
To date, definite depiction of anatomy or pathologies of bony structures requires ionizing radiation by using radiographs or computed tomography (CT) since conventional magnetic resonance imaging (MRI) that does not require ionizing radiation cannot depict bony structures well. Modern MR techniques, collectively referred to as ultrashort time to echo (UTE) sequences, have overcome this issue by acquiring the signal data much faster and therefore are able to acquire sufficient MR signal from bony structures. The investigators want to investigate if UTE sequences are capable to depict bony anatomy and pathology similar to imaging examination techniques involving ionizing radiation. Healthy adult and minor participants, as well as adult and minor participants, referred for a clinically indicated MRI involving the skeletal system will be included.

ELIGIBILITY:
Inclusion criteria:

* adults and minors (all ages) capable of giving informed consent or have a legal representative capable of giving consent on the participant's behalf. Informed Consent as documented by signature (Appendix Informed Consent Form)
* for participants referred for a clinical indicated MRI (primary objective) inclusion criterion is the presence of radiographs or a CT scan of the part of the skeletal system that is under investigation within the clinical indicated MRI
* for healthy volunteers (secondary objective) any volunteer that is not referred for a clinical indicated MRI scan

Exclusion criteria:

* women who are pregnant
* general known contraindications for MRI (e.g., non-MR compatible pacemaker)
* homeless persons, or persons with active drug/alcohol dependence or abuse history

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the accuracy of bone anatomy size dimensions measurements between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 1 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be:
  - size dimensions of the bony structures in three dimensions in millimeter
Comparison of the accuracy of cortical bone depiction between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 2 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be
  - clearly visibility of the cortical bone according to a scale 1-4 (1 = cortical bone not good visible; 4 = cortical bone good visible)
Comparison of the accuracy of cancellous bone depiction between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 3 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be
  - clearly visibility of the cancellous bone according to a scale 1-4 (1 = cancellous bone not good visible; 4 = cancellous bone good visible)
Comparison of the accuracy of calcification depiction between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 4 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be
  - clearly visibility of calcifications according to a scale 1-4 (1 = calcification not good visible; 4 = calcification good visible)
Comparison of the diagnostic performance for depiction of bony anatomy between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 5 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be:
  - diagnostic performance measurements for the depiction of bony anatomy (sensitivity, specificity, accuracy)
Comparison of the diagnostic confidence for depiction of bony anatomy between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 5 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be:
  - diagnostic confidence measurements for the depiction of bony anatomy (1-4, 1=anatomical bony structure certainly absent, 4= certainly present)
Comparison of the Signal-to-noise (SNR) measurements between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 6 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be:
  - Signal-to-noise (SNR)
Comparison of the Contrast-to-noise (CNR) measurements between regular MRI and UTE MRI | There is no baseline and follow-up examination for this study. The outcome measure will be assessed on the same day after the MRI examination is finished.
  Outcome measure 7 will be to compare the bone anatomy as visible on the radiation-free UTE images with the reference standard (pre-existing radiographs or CT) during readouts performed by radiologists. The measurements for the primary endpoint will specifically be:
  - Contrast-to-noise (CNR)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Guggenberger, MD, PD, Principal Investigator — Universitätsspital Zürich; Christian Kellenberger, MD, Principal Investigator — Kinderspital Zürich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No